CLINICAL TRIAL: NCT06413875
Title: The Effect of Menopausal Symptoms Specific Education Given to Women in Menopause Via WhatsApp on Quality of Life and Genital Self-Image
Brief Title: Effectiveness of Education Specific to Menopause Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bartın Unıversity (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Ebru Cirban Ekrem, Lecturer, Bartın Unıversity
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: makale
Record Dates: First submitted 2024-05-07; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Menopause
Keywords: Genital image; menopause; woman; symptom; quality of life
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The population of the study, which has a classical experimental design with a pretest-posttest control group, was comprised of women between the ages of 45-65 across Turkey. According to the power analysis performed in the G*Power3.1 Program, the sample size was calculated as 64 participants for each group, with an effect size (0.418), 95% power and 0.05 type 1 error, and was completed with 158 women. Data were collected with the Introductory Information Form, the Menopause-Specific Quality of Life Scale (MSQLS) and the Female Genital Self-Image Scale (FGSIS). The research was conducted online via WhastApp in a pretest-educational intervention-posttest design. The data were analyzed in the SPSS 26.0 package program.
Who Masked: Participant
Masking Description: Participants were informed about the research, and then participants who agreed to participate in the research were given a number respectively. After the targeted sample number was reached, all participants were divided into intervention and control groups using a simple random numbers table.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- enterprise group (Experimental): The data collection form was sent online to the participants in the sample and they were asked to fill it out (pre-test). Two separate groups were opened on WhatsApp for the intervention and control groups. For this reason, in this study, the educational intervention included sending an informative video once a week and informative messages three days a week for four weeks.In the intervention part of the study, after all participants filled out the data collection form, the intervention group was informed about Menopause once a week on the first day of each week for four weeks. An information video prepared in line with the topics specified in the Symptom-Specific Training Booklet has been sent. Informative messages were sent via WhatsApp three days a week, in parallel with the training topic of each week (training intervention).After the training, a data collection form was sent to the intervention group via WhatsApp and the participants were asked to fill it out again (posttest).
  Interventions: Other: education
- control group (No Intervention): The data collection form was sent online to the participants in the sample and they were asked to fill it out (pre-test). No educational intervention was given to the control group. After the training, a data collection form was sent to the control group via WhatsApp and the participants were asked to fill it out again (posttest).

INTERVENTIONS:
Other: education — Education Specific to Menopause Symptoms
  Arms: enterprise group

SUMMARY:
Objective: To determine the effect of menopausal symptom-specific education given to menopausal women via WhatsApp on their quality of life and genital self-image.

Methods: The population of the study, which has a classical experimental design with a pretest-posttest control group, was comprised of women between the ages of 45-65 across Turkey. According to the power analysis performed in the G*Power3.1 Program, the sample size was calculated as 64 participants for each group, with an effect size (0.418), 95% power and 0.05 type 1 error, and was completed with 158 women. Data were collected with the Introductory Information Form, the Menopause-Specific Quality of Life Scale (MSQLS) and the Female Genital Self-Image Scale (FGSIS). The research was conducted online via WhastApp in a pretest-educational intervention-posttest design. The data were analyzed in the SPSS 26.0 package program.

DETAILED DESCRIPTION:
Objective: To determine the effect of menopausal symptom-specific education given to menopausal women via WhatsApp on their quality of life and genital self-image.

Methods: The population of the study, which has a classical experimental design with a pretest-posttest control group, was comprised of women between the ages of 45-65 across Turkey. According to the power analysis performed in the G*Power3.1 Program, the sample size was calculated as 64 participants for each group, with an effect size (0.418), 95% power and 0.05 type 1 error, and was completed with 158 women. Data were collected with the Introductory Information Form, the Menopause-Specific Quality of Life Scale (MSQLS) and the Female Genital Self-Image Scale (FGSIS). The research was conducted online via WhatsApp between April and December 2023, using the snowball sampling method with participants who met the inclusion criteria. In snowball sampling, first of all, contact was made with one of the units of the universe. With the help of the contacted unit, a third unit was contacted. In this way, the sample size expanded like a snowball growing. First, the participants around the researchers were reached, and then the participants' circle was reached. The data collection form was sent online to the participants in the sample and they were asked to fill it out (pre-test). Two separate groups were opened on WhatsApp for the intervention and control groups. It has been stated in the literature that video and informative message interventions performed three days a week for 3-6 weeks are effective. For this reason, in this study, the educational intervention included sending an informative video once a week and informative messages three days a week for four weeks.18,19 In the intervention part of the study, after all participants filled out the data collection form, the intervention group was informed about Menopause once a week on the first day of each week for four weeks. An information video prepared in line with the topics specified in the Symptom-Specific Training Booklet has been sent. Informative messages were sent via WhatsApp three days a week, in parallel with the training topic of each week (training intervention). No educational intervention was given to the control group. After the training, a data collection form was sent to both the intervention and control groups via WhatsApp and the participants were asked to fill it out again (posttest). After the final test phase of the research was completed, training videos and informative messages were sent to the participants in the control group via WhatsApp. The data collection form was filled out using the self-report method in approximately 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 45-65 between April and December 2023,
* in the pre/peri/postmenopausal period,
* not receiving hormone replacement therapy in the last 6 months,
* not having had a gynecological operation,
* women who have internet access, (6) use a smartphone,
* voluntarily agree to participate in the study.

Exclusion Criteria:

* Those who filled out the data collection form incompletely

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Menopausal women between the ages of 45-65
Enrollment: 158 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
The total quality of life scale score of the intervention group that received training on menopause symptoms was better than the control group. | 4 weeks
  Education Specific to Menopause Symptoms
The genital self-image scale total score of the intervention group that received training on menopause symptoms was better than the control group. | 4 weeks
  Education Specific to Menopause Symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Ebru Cirban Ekrem, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The research is in the article writing phase. It will be published as an article.